CLINICAL TRIAL: NCT05148663
Title: CCMs Among Hispanic Population Study Group (CHIPS)
Brief Title: CCM Blood Biomarker Validation Study
Status: Terminated | Type: Observational
Why Stopped: Leaving the institution
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Jun Zhang, Ph.D., ScD, Associate Professor, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E21010
Record Dates: First submitted 2021-07-27; First posted 2021-12-08 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hemorrhagic Stroke, Intracerebral; Cerebral Cavernous Malformation
MeSH Terms: conditions — Hemorrhagic Stroke; Hemangioma, Cavernous, Central Nervous System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma can be used to isolated human DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- blood drawing and hemorrhagic events in CCM patients: planned for three blood drawing before surgery
  Interventions: Diagnostic Test: CCM Hemorrhagic Panel
- blood drawing for age/gender/ethnicity matched controls: Blood draw from Control patients with no inflammation
  Interventions: Diagnostic Test: CCM Hemorrhagic Panel

INTERVENTIONS:
Diagnostic Test: CCM Hemorrhagic Panel — Biomarker

SUMMARY:
Cerebral cavernous malformations (CCMs), one of the most common microvascular malformations in the capillary beds of the brain, are susceptible to hemorrhagic stroke. As an autosomal dominant disorder with incomplete penetrance, the majority of CCM gene mutation carriers are largely asymptomatic but when symptoms occur, the disease has typically reached the stage of focal hemorrhage with irreversible brain damage. Currently, the invasive neurosurgery removal of CCM lesions is the only treatment option, despite the recurrence of the symptoms after surgery. Therefore, there is a grave need for prognostic/monitoring biomarkers as risk predictors for stroke prevention. The objective of the proposal is to develop a set of blood prognostic/monitoring biomarkers as precise risk indicators for stroke prevention. In this project, the plan is to validate the novel serum biomarkers identified in Ccms animal models and human CCMs patients, and utilize these biomarkers with statistical algorithms for risk prediction of hemorrhagic CCMs. This proposal has been formulated based on recent findings of five serum etiological biomarkers associated with disruption of the Blood-Brain Barrier (BBB), the first step for hemorrhagic CCMs in Ccm mice models. This work will lay the groundwork for larger human trials for final validation and revolutionary potential clinical applications.

DETAILED DESCRIPTION:
Cerebral cavernous malformations (CCMs), one of the most common vascular malformations, are characterized by abnormally dilated intracranial capillaries resulting in increased susceptibility to hemorrhagic stroke. As an autosomal dominant disorder with incomplete penetrance, the majority of CCMs gene mutation carriers are largely asymptomatic but when symptoms occur, the disease has typically reached the stage of focal hemorrhage with irreversible brain damage. Currently, the invasive neurosurgery removal of CCM lesions is the only treatment option, despite the recurrence of symptoms after surgery. Therefore, there is a grave need for prognostic/monitoring biomarkers as risk predictors for stroke prevention. The goal is to develop a set of blood prognostic biomarkers as risk predictors for stroke prevention. The objective of this project is to validate novel serum biomarkers identified in Ccm animal models in human blood that could predict the risk of hemorrhagic events. The central hypothesis is that quantitative detection of certain serum biomarkers can be utilized to predict the timing of hemorrhagic events. The hypothesis has been formulated based on the recent findings of five serum etiological biomarkers associated with disruption of the Blood-Brain Barrier (BBB), which could lead to hemorrhagic events. Taking advantage of the research team's expertise in Ccm pathology and serum biomarkers, the central hypothesis will be tested to achieve the study goal by pursuing the following three revolutionary aims in two phases, starting from the phase 1 with the first two biomarker discovery aims (1, 2):

1. Validate blood prognostic/monitoring biomarkers with the optimized detection platform for hemorrhagic stroke prevention. The working hypothesis is that expression levels of certain blood molecules are correlated with the progression of a disrupted BBB. In this aim, serum biomarkers identified in Ccms mice will be validated in the blood samples of CCM patients to evaluate their feasibility and reliability. The correlation functions between the serum/plasma levels of biomarkers and the progression of a disrupted BBB identified in Ccms mice will be tested using the "gold standard", enzyme-linked immunosorbent assay (ELISA) platform in CCM patients for 1a). Clinical preparation for large cohort CCM analysis; 1b). Validating serum progesterone (PRG) as a biomarker, and 1c). Validating 4 etiological serum peptide biomarkers with the optimized ELISA platform in CCM patients.
2. To optimize the sensitivity, specificity, dynamic range, and reliability of biomarkers using the cutting-edge multiplex platform to predict risks of hemorrhagic stroke. The working hypothesis is that the measurement parameters of blood biomarkers, such as sensitivity, specificity, dynamic working range, and inter/intra variability, can be drastically improved with a larger sample size, improved clinical definitions, and better detection platforms. High-performance ELISAs will be continuously utilized for validating etiological biomarkers. To ensure the highest sensitivity and specificity, a robust automatic multiplex platform for the repetitive analysis of large cohorts is essential to validate biomarkers for hemorrhagic strokes. Linear or logistic regression analysis will be performed to delineate the correlation between validated biomarkers and those of clinical criteria. In this aim, the will 2a). Improve sensitivity and specificity of candidate blood biomarkers through correlation equations were optimized with increased CCM blood sample sizes and updated clinical information; 2b). Define new biomarkers using high-throughput omic approaches, and 2c). Improve sensitivity and increase dynamic working range of blood biomarkers with a multiplex bead array assay (MBAA) platform and optimized protocols.

Phase-2 Aim: 3) Improve clinical utility of validated prognostic/monitoring biomarkers with optimized algorithms in larger cohorts in preparation for human clinical trials. The working hypothesis is that clinical sensitivity and specificity of blood biomarkers can be further improved through a blindly test-retest approach in larger independent human cohorts. This aim will provide sufficient proof that the clinical utility of blood biomarkers can be improved and utilized to predict the risk of hemorrhagic stroke, laying the groundwork for future clinical trials and possible future revolutionary clinical applications. The research team will continue to 3a). Improve clinical utility by optimizing the precision of prognostic/monitoring algorithms of validated biomarker(s)/panel(s) using larger cohorts; 3b). Further improve clinical utility by confirming reliability of validated biomarker(s)/panel(s) in a larger cohort; and 3c). Confirm validated prognostic/monitoring biomarker(s)/panel(s) are ready for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. 10 to 78 years of age.
2. Medical history meets the criteria for the International Classification of Diseases diagnosis codes 10 (ICD-10) for cerebral cavernous malformations (CCMs) (Q28.3) or stroke/epilepsy.
3. Has a family member whose medical history meets the criteria for the International Classification of Diseases diagnosis codes for cerebral cavernous malformations (CCMs) (Q28.3) or stroke/epilepsy.
4. Has a relatively complete medical history that can be accurately confirmed by an interview or electronic and/or paper medical records.
5. Hispanic and non-Hispanic Americans.

Exclusion Criteria:

N/A

Ages: 10 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mexican Hispanic population
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Identification and validation of at least (>1) biomarker(s) with a significant p-value (p≤ 0.001) to correlate with the progression of hemorrhagic events in CCM patients using our optimized ELISAs. | the first two years
  Confirmation of at least (>1) biomarker(s) is essential for the feasibility assessment of this project after three years investigation and validation in the mid-sized cohorts (~300 each cases/controls). Thus, to assess the consistency of the measurement between different CCM cohorts at the end of the 1st phase, the blinded test-retest reliability (r2) will be calculated with a relatively strong outcome range (~0.65-0.70, p=0.005) on at least (>1) positively/negatively correlated biomarker(s).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Principal Investigator — TTUHSC
Locations (1):
- TTUHSC El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT05148663/Prot_000.pdf
  • Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT05148663/ICF_001.pdf